CLINICAL TRIAL: NCT02722200
Title: Investigating the Central and Peripheral Mechanisms by Which Glucocorticoids Affect Hunger
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1510016716; 2R01DK020495-42 (NIH)
Record Dates: First submitted 2016-03-22; First posted 2016-03-29 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Obesity
Keywords: fMRI obesity
MeSH Terms: conditions — Obesity | interventions — Hydrocortisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous glucocorticoids (Experimental): Subjects in the glucocorticoids arm will receive an infusion of hydrocortisone overnight in the research unit prior to fMRI testing on either the first or second visit.
  Interventions: Drug: hydrocortisone
- Intravenous saline (Placebo Comparator): Subjects in the saline arm will receive an infusion of saline overnight in the research unit prior to fMRI testing on either the first or second visit.
  Interventions: Other: saline

INTERVENTIONS:
Drug: hydrocortisone — Hydrocortisone will be used as the steroid of choice because it is bio-identical to cortisol and is subject to the same metabolism as cortisol.
  Arms: Intravenous glucocorticoids
Other: saline — Saline will be used as the placebo comparator. It will be administered in the same manner as the active drug.
  Arms: Intravenous saline

SUMMARY:
The purpose of this study is to examine if glucocorticoids will change neural activation in regions of the corticolimbic-striatal system that regulate feeding.

DETAILED DESCRIPTION:
The primary hypothesis tested in this study will be to determine if that in response to food cues, glucocorticoids will change neural activation in regions of the corticolimbic-striatal system that regulate feeding. It is anticipate that these changes will correlate with hunger ratings and food intake. Further, this research will also examine if glucocorticoids will increase the basal metabolic rate and alter multiple systemic appetite-regulating hormones compared to saline. It is expected that these changes will correlate positively with hunger ratings and food intake as well.

ELIGIBILITY:
Inclusion Criteria:

* BMI < = 26 kg/m2
* Ability to read and write English

Exclusion Criteria:

* Creatinine > 1.5
* Hgb < 10 mg/dL
* ALT > 2.5 x ULN
* Untreated thyroid disease
* Uncontrolled or severe hypertension
* Known neurological disorders
* Diabetes or impaired glucose tolerance
* Untreated or severe psychiatric disorders
* Malignancy
* Endogenous hypercortisolism
* Addison's disease
* Bleeding disorders
* Smoking
* Current or recent steroid use in the last 3 months
* Illicit drug use
* Eating disorders
* Drug or alcohol addiction
* History of claustrophobia
* Pregnancy
* Breastfeeding
* Contraindications to MRI
* Use of any psychoactive medication within the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Change in Brain Response to Food Imagery | 90 minutes
  Brain response to images of food either during hydrocortisone infusion or saline infusion will be measured through fMRI. Brain response is operationally defined as the change in functional MRI-measured blood oxygen levels in specific regions of the brain between the resting state and intervention state. The fMRI sequences last anywhere from 1-5 min. Total scan time will be approximately 90 minutes. The slices taken with each sequences equal 25-75.
  The outcome is a comparison between the resting oxygen levels and oxygen levels during the interventions. BioImage Suite software is used to categorize if there is a significance between the two levels at a p < 0.05.
Average Hunger Rating | 90 minutes
  Average hunger rating will be captured using the Visual Food Cue Task. This standardized method presents a series of images consisting of high calorie food, low calorie food, and non-food pictures presented randomly across four runs during the fMRI session. Each picture will be presented only once in a randomized order for each participant.
  Participants will be instructed to rate their "hunger", "liking" and "wanting" of the item on a 9-point Likert scale utilizing a 4-key button box. The hunger, wanting, and liking scales are all rated on a scale of 1-9, 1 being the least and 9 being the most. These scores are presented as an average across measurement points during the fMRI. Every time a food image is shown, the rater provides a rating of hunger, wanting and liking of it- people will be shown approximately 40-60 photos.

SECONDARY OUTCOMES:
Average Wanting Rating | 90 minutes
  Average wanting rating will be captured using the Visual Food Cue Task. This standardized method presents a series of images consisting of high calorie food, low calorie food, and non-food pictures presented randomly across four runs during the fMRI session. Each picture will be presented only once in a randomized order for each participant. Participants will be instructed to rate their "hunger", "liking" and "wanting" of the item on a 9-point Likert scale utilizing a 4-key button box. The hunger, wanting, and liking scales are all rated on a scale of 1-9, 1 being the least and 9 being the most. These scores are presented as an average across measurement points during the fMRI.
Average Liking Rating | 90 minutes
  Average wanting rating will be captured using the Visual Food Cue Task. This standardized method presents a series of images consisting of high calorie food, low calorie food, and non-food pictures presented randomly across four runs during the fMRI session. Each picture will be presented only once in a randomized order for each participant. Participants will be instructed to rate their "hunger", "liking" and "wanting" of the item on a 9-point Likert scale utilizing a 4-key button box. The hunger, wanting, and liking scales are all rated on a scale of 1-9, 1 being the least and 9 being the most. These scores are presented as an average across measurement points during the fMRI.
Total Cortisol | Baseline
  Total cortisol will be collected from serum at the beginning and end of the procedure.
Total Cortisol | 90 minutes
  Total cortisol will be collected from serum at the beginning and end of the procedure.
Free Cortisol | Baseline
  Free cortisol will be collected from serum at the beginning and end of the procedure.
Free Cortisol | 90 minutes
  Free cortisol will be collected from serum at the beginning and end of the procedure.
Cortisone | Baseline
  Cortisone will be collected from serum at the beginning and end of the procedure.
Cortisone | 90 minutes
  Cortisone will be collected from serum at the beginning and end of the procedure.
Adrenocorticotropic Hormone | Baseline
  Adrenocorticotropic Hormone (ACTH) will be collected from serum at the beginning and end of the procedure.
Adrenocorticotropic Hormone | 90 minutes
  Adrenocorticotropic Hormone (ACTH) will be collected from serum at the beginning and end of the procedure.
Glucose | Baseline
  Glucose will be collected from serum at the beginning and end of the procedure.
Glucose | 90 minutes
  Glucose will be collected from serum at the beginning and end of the procedure.
Glucagon | Baseline
  Glucagon will be collected from serum at the beginning and end of the procedure.
Glucagon | 90 minutes
  Glucagon will be collected from serum at the beginning and end of the procedure.
Insulin | Baseline
  Insulin will be collected from serum at the beginning and end of the procedure.
Insulin | 90 minutes
  Insulin will be collected from serum at the beginning and end of the procedure.
Leptin | Baseline
  Leptin will be collected from serum at the beginning and end of the procedure.
Leptin | 90 minutes
  Leptin will be collected from serum at the beginning and end of the procedure.
Ghrelin | Baseline
  Ghrelin will be collected from serum at the beginning and end of the procedure.
Ghrelin | 90 minutes
  Ghrelin will be collected from serum at the beginning and end of the procedure.
Neuropeptide Y | Baseline
  Neuropeptide Y (NPY) will be collected from serum at the beginning and end of the procedure.
Neuropeptide Y | 90 minutes
  Neuropeptide Y (NPY) will be collected from serum at the beginning and end of the procedure.
Glucagon-like peptide-1 | Baseline
  Glucagon-like peptide-1 (GLP-1) will be collected from serum at the beginning and end of the procedure.
Glucagon-like peptide-1 | 90 minutes
  Glucagon-like peptide-1 (GLP-1) will be collected from serum at the beginning and end of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided